CLINICAL TRIAL: NCT01048125
Title: Characterization of Sympathetic Nerve Activity in Stress Cardiomyopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty in recruitment and resource restraints
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Anand Chockalingam, Professor, Cardiology, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1141858
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Cardiomyopathy
Keywords: Stress-induced cardiomyopathy; Takotsubo cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Takotsubo Cardiomyopathy | interventions — Nitroprusside; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Subjects with documented stress cardiomyopathy who would serve as the study group. Sympathetic Nerve Activity; Mental StrCold Pressor Testess Test (Color Word Test); The Modified Oxford Technique for Baroreflex Sensitivity; Cold Pressor Test; Echocardiographic evaluation
  Interventions: Device: Sympathetic Nerve Activity; Behavioral: Mental Stress Test (Color Word Test); Drug: The Modified Oxford Technique for Baroreflex Sensitivity; Other: Cold Pressor Test; Device: Echocardiographic evaluation
- Control (Active Comparator): Control subjects will be age and sex matched otherwise healthy people with no prior cardiac disease or other severe medical conditions. Sympathetic Nerve Activity; Mental Stress Test (Color Word Test); The Modified Oxford Technique for Baroreflex Sensitivity; Cold Pressor Test; Echocardiographic evaluation
  Interventions: Device: Sympathetic Nerve Activity; Behavioral: Mental Stress Test (Color Word Test); Drug: The Modified Oxford Technique for Baroreflex Sensitivity; Other: Cold Pressor Test; Device: Echocardiographic evaluation

INTERVENTIONS:
Device: Sympathetic Nerve Activity — Resting Sympathetic Nerve Activity
Behavioral: Mental Stress Test (Color Word Test) — A printed word will be shown to the subject, displayed in a color different from the color it actually names. The subject will be asked to say the color that the word is printed in as quickly as possible. For example if the word "green" is written in blue ink, they will say "blue." This mental stress procedure will be used to cause brief changes in heart rate and blood pressure.
Drug: The Modified Oxford Technique for Baroreflex Sensitivity — Sodium nitroprusside (100 µg) will be infused intravenously as a bolus, followed 60 seconds later by a bolus of phenylephrine hydrochloride (150 µg). Infusion of nitroprusside will decrease blood pressure approximately 10-15 mmHg below baseline values. Subsequent phenylephrine infusion will increase blood pressure approximately 10-15 mmHg above baseline values. Nitroprusside and phenylephrine have been used extensively to assess baroreflex sensitivity in healthy as well as heart failure populations. Additionally, the dosages being used have been shown to minimize the risk of excessive decreases or increases in blood pressure.
  Other Names: Sodium Nitroprusside; Phenylephrine hydrochloride
Other: Cold Pressor Test — The subject will be asked to place their hand in ice water for 2 minutes. This procedure will be used to cause transient changes in sympathetic nerve activity, heart rate and blood pressure.
Device: Echocardiographic evaluation — Transthoracic echocardiography with 2D, color and pulse Doppler will be employed in all of our subjects. Baseline left ventricular function, systolic as well as diastolic, will be quantified.

SUMMARY:
Stress (Takotsubo) cardiomyopathy (SC) is a peculiar form of acute, reversible myocardial dysfunction predominantly affecting the apical and mid left ventricular segments.

In this institution over the last two to three years the investigators have identified more than a dozen patients with stress cardiomyopathy. The investigators' overarching goal is to characterize these individuals with the hope of identifying risk factors and developing strategies to prevent the occurrence of SC in situations where the likelihood in susceptible individuals may be high.

DETAILED DESCRIPTION:
Stress (Takotsubo) cardiomyopathy (SC) is a peculiar form of acute, reversible myocardial dysfunction predominantly affecting the apical and mid left ventricular segments. This was originally described in Japan but is increasingly recognized all over the world especially in older women. There is evidence to support that excess sympathetic activation and catecholamine surges are potential mechanisms that cause this temporary myocardial 'stunning'. The amount of catecholamines in circulation of patients with SC was 2 to 3-fold higher when compared to subjects with acute myocardial infarction related equivalent cardiac dysfunction [Wittstein, et al. NEJM, 2005].

In this institution over the last two to three years the investigators have identified more than a dozen patients with stress cardiomyopathy. This diagnosis has been confirmed by echocardiographic documentation of normalization of left ventricular function over a course of few days to weeks. The investigators' overarching goal is to further characterize these individuals with the hope of identifying risk factors and developing strategies to prevent the occurrence of SC in situations where the likelihood in susceptible individuals may be high.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stress cardiomyopathy in the past

Exclusion Criteria:

* Coronary artery disease (CAD), primary coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Cardiac dysfunction
* Heart failure
* Significant arrhythmias
* Severe chronic obstructive pulmonary disease (COPD)
* Diabetic neuropathy
* Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Chockalingam, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were consented, but due to difficulty in recruitment and resource restraints the study did not progress as expected and was closed.
Groups:
- Control: Control subjects will be age and sex matched otherwise healthy people with no prior cardiac disease or other severe medical conditions. Sympathetic Nerve Activity; Mental Stress Test (Color Word Test); The Modified Oxford Technique for Baroreflex Sensitivity; Cold Pressor Test; Echocardiographic evaluation
  Sympathetic Nerve Activity: Resting Sympathetic Nerve Activity
  Mental Stress Test (Color Word Test): A printed word will be shown to the subject, displayed in a color different from the color it actually names. The subject will be asked to say the color that the word is printed in as quickly as possible. For example if the word "green" is written in blue ink, they will say "blue." This mental stress procedure will be used to cause brief changes in heart rate and blood pressure.
  The Modified Oxford Technique for Baroreflex Sensitivity: Sodium nitroprusside (100 µg) will be infused intravenously as a bolus, followed 60 seconds later by a bolus of phenylephrine hydrochloride
Period: Overall Study
Arm/Group | Study Group | Control
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to difficulty in recruitment and resource restraints the study did not progress as expected and was closed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
  <=18 years |  |  | 0
  Between 18 and 65 years |  |  | 0
  >=65 years |  |  | 0
Gender
  Female |  |  | 0
  Male |  |  | 0
Region of Enrollment
  United States |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Identifying Risk Factors and Developing Strategies to Prevent the Occurrence of Stress Cardiomyopathy in Situations Where the Likelihood in Susceptible Individuals May be High.
Time Frame: 2 years
Population: Due to difficulty in recruitment and resource restraints the study did not progress as expected and was closed.
Arm/Group | Study Group | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Study Group | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
2 participants were consented, but due to difficulty in recruitment and resource restraints the study did not progress as expected and was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes